CLINICAL TRIAL: NCT02657187
Title: The Neuromuscular Effect of Rocuronium in Patient Measuring Muscle Mass by Bioelectrical Impedance Analysis
Brief Title: The Neuromuscular Effect of Rocuronium in Patient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Go Eun Bae (Other)
Responsible Party: Sponsor-Investigator, Go Eun Bae, Clinical instructor, Korea University Anam Hospital
Organization: Korea University Anam Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Inbody2
Record Dates: First submitted 2016-01-13; First posted 2016-01-15 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Anesthesia
MeSH Terms: interventions — Rocuronium

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- rocuronium 1 (Experimental): Participant measure muscle mass by bioelectrical impedance analysis (Inbody 720, Inbody, Seoul, Korea) and the dose of rocuronium is 0.24mg per muscle mass(kg).
  Interventions: Device: Inbody; Drug: Rocuronium
- rocuronium 2 (Experimental): Participant measure muscle mass by bioelectrical impedance analysis (Inbody 720, Inbody, Seoul, Korea) and the dose of rocuronium is 0.32mg per muscle mass(kg).
  Interventions: Device: Inbody; Drug: Rocuronium
- rocuronium 3 (Experimental): Participant measure muscle mass by bioelectrical impedance analysis (Inbody 720, Inbody, Seoul, Korea) and the dose of rocuronium is 0.40mg per muscle mass(kg).
  Interventions: Device: Inbody; Drug: Rocuronium
- rocuronium 4 (Experimental): Participant measure muscle mass by bioelectrical impedance analysis (Inbody 720, Inbody, Seoul, Korea) and the dose of rocuronium is 0.48mg per muscle mass(kg).
  Interventions: Device: Inbody; Drug: Rocuronium

INTERVENTIONS:
Device: Inbody — Participant measure muscle mass by bioelectrical impedance analysis (Inbody 720, Inbody, Seoul, Korea) after fast for eight hours.
Drug: Rocuronium — The individual dose method was used for the determination of the dose response of rocuronium. After induction of anesthesia, four groups of 40 patients each received randomly one of the four doses of rocuronium ( 0.24, 0.32, 0.40, 0.48mg/muscle mass(kg))
  Other Names: Esmeron(MSD Korea Ltd.)

SUMMARY:
Rocuronium block neuromuscular transmission at the neuromuscular junction, causing paralysis of the affected skeletal muscles. There have been several studies reported positive relationship between muscle mass and amount of neuromuscular junction. The purpose of this study is to find 50% effective dose and 95% effective dose of rocuronium according to muscle mass.

DETAILED DESCRIPTION:
Rocuronium block neuromuscular transmission at the neuromuscular junction, causing paralysis of the affected skeletal muscles. There have been several studies reported positive relationship between muscle mass and amount of neuromuscular junction. Until now, dose of rocuronium has been judged by patient's weight and height. When the rocuronium was developed, 50% effective dose and 95% effective dose of rocuronium was calculated by patient corrected body weight which used weight and height. However, height and weight do not represent exact muscle mass. The purpose of this study is to find 50% effective dose and 95% effective dose of rocuronium according to muscle mass. Measurement of muscle mass will be obtained using bioelectrical impedence analysis.

ELIGIBILITY:
Inclusion Criteria:

* All patient who undergo general anesthesia

Exclusion Criteria:

* Liver and kidney disease
* Any types of muscle disorder.
* Metal materials or pacemaker in body

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-07 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
percentage of neuromuscular block | ten minutes
  percentage of neuromuscular block is calculated by ratio of T1 to T4. T1 is result of first stimulation and T4 is result of fourth stimulation which are obtained by commonly used neuromuscular monitoring device.

SECONDARY OUTCOMES:
onset time | ten minutes
  time from the end of injection of rocuronium until the maximal depression of T1 which is result of first twitch

OTHER OUTCOMES:
lag time | ten minutes
  time from the end of injection of rocuronium until the first depression of the twitch response

CONTACTS AND LOCATIONS:
Overall Officials: Go eun Bae, M.D., Study Director — Korea University Anam Hospital
Locations (1):
- Korea university anam hospital, Seoul, South Korea